CLINICAL TRIAL: NCT03921762
Title: Comparison of Visual Outcomes After Bilateral Implantation of a New Extended Depth of Focus (EDOF) IOL Twinset With Bilateral Standard EDOF IOLs
Brief Title: Comparison of a New EDOF-IOL With a Standard-EDOF-IOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Principal Investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Artis Active
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Cataract
Keywords: Cataract surgery; Enhanced depth of focus (EDOF); Intraocular lens
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Artis Active IOL (Experimental): Artis Active IOLs (Artis Active Mid, Artis Active Plus) will be implanted in patients eyes during cataract surgery
  Interventions: Procedure: Cataract surgery with Artis Active IOLs
- AT Lara IOL (Experimental): AT Lara IOLs will be implanted in patients eyes during cataract surgery
  Interventions: Procedure: Cataract surgery with AT Lara IOLs

INTERVENTIONS:
Procedure: Cataract surgery with Artis Active IOLs — Patients will be implanted with the Artis Active IOLs during cataract surgery
  Arms: Artis Active IOL
Procedure: Cataract surgery with AT Lara IOLs — Patients will be implanted with the AT Lara IOLs during cataract surgery
  Arms: AT Lara IOL

SUMMARY:
Comparison of the new extended depth of focus (EDOF) intraocular lens (IOL) ARTIS ACTIVE, which is designed as a twinset of IOLs, with the standard EDOF IOL AT Lara .

DETAILED DESCRIPTION:
Spectacle independence is a central aim in modern cataract surgery. Although bilateral monofocal IOL implantation, aiming for emmetropia or low myopia, leads to high levels of patient satisfaction in distance vision, spectacle dependence for reading and other near vision tasks is the usual result.

The option commonly used to achieve spectacle independence are multifocal intraocular lenses (IOLs). Multifocal IOLs either use a refractive or diffractive design or a combination of both or segmented asymmetric optics. The principal of the refractive design is based on changing the route of light rays by thickness, curvature and optical density of the lens. The principal of diffractive design is based on scattering of light rays when passing an edge in the material of the lens. Usually, the characteristic diffractive ring patterns are incorporated on the posterior surface of an IOL, whereas the anterior lens surface remains purely refractive. One potentially negative aspect of multifocal refractive IOLs is pupil size dependence, another is loss of light energy to higher order diffraction which is not useful for the patient. In clinical studies, diffractive lenses resulted in a better outcome in terms of optical quality, better contrast sensitivity, and less photic phenomena (dysphotopsia such as halos and glare) compared to refractive lenses.

Until recently multifocal lenses were typically bifocal with a focus assigned to near and a focus assigned to far vision. However, the intermediate working distance is poorly covered by the bifocal design. Since objects commonly viewed in this distance include computer displays and tablets, the intermediate distance has become a crucial part in daily life. Variations in the addition of power chosen for near vision provided some intermediate visual acuity, but still suboptimal. Therefore, a new concept of multifocality has been introduced, the trifocal lens. Trifocal IOLs provide three focal distances: far, intermediate, and near. This ideally results in even less spectacle dependence, including for computer work. However, one potential disadvantage of trifocal IOLs is slightly poorer near vision compared to bifocal IOLs with need for reading glasses for prolonged fine near work and loss of contrast sensitivity in the intermediate distance.

A better intermediate performance concerning contrast vision compared to trifocal IOLs can be reached using enhanced depth of focus (EDOF) lenses. These IOLs have an extended far focus area which reaches to the intermediate distance, providing high-quality vision over a continuous range of focus, rather than distinct foci with blur in between.

To provide similar outcomes to trifocal IOLs, mix-and-match of additions ("blended vision") is another option, in which additions of multifocal IOLs between both eyes differ. The idea behind it is to improve the contrast in the intermediate distance compared to trifocal IOLs. The combination of +1.75D/ +4D10 and +1.5D/ +3D11 successfully achieved a regular defocus curve, but patient's subjective binocular comfort was not determined. To preserve the binocular balance between the eyes, a difference in addition of 0.5D was proposed and the combination of +2.5D/ +3D showed similar results as trifocal IOLs, except in the intermediate range of -1D and -1.5D.

Therefore, it would be necessary to provide an IOL with a continuum of good visual acuity from distance to 40 cm using binocularity to preserve binocular balance between the eyes. Hence, the primary objective of this study is to compare a new designed twinset of EDOF IOLs, ARTIS ACTIVE (Artis Active Mid and Artis Active Plus), with the standard EDOF IOL AT Lara in binocular visual acuity at 40 cm. Secondary objective is to compare binocular contrast sensitivity (with and without glare), binocular defocus curves with distance correction, monocular and binocular halos, and reading speed between the two IOLs.

ELIGIBILITY:
Inclusion Criteria:

* > 50 years old
* Bilateral age-related cataract
* Qualify for bilateral implantation within 1 month
* No previous refractive or ocular surgery
* Available IOL dioptre range: 18 to 27D
* Expected postoperative astigmatism ≤ 0.75D

Exclusion Criteria:

* Pupil > 4 mm
* Occupation requiring night-time driving or any occupation incompatible with multifocality
* Acute or chronic disease or illness that would increase risk or confound study results [e.g. diabetes mellitus (with retinopathy), immunocompromised, glaucoma, epiretinal membrane, cornea guttata, etc….] found to be relevant by the investigators
* Amblyopia, strabismus
* Extremely shallow anterior chamber
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome, uveitis, Marfan's syndrome)
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic/ scotopic conditions)
* Instability to place the intraocular lens safely at the location planned
* Pregnancy (pregnancy test will be taken pre-operatively in women of reproductive age)

Ages: 50 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2018-10-29 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of binocular near visual acuity | 12 months
  Binocular near visual acuity in logMar will be measured at 40 cm distance using an ETDRS visual acuity chart

SECONDARY OUTCOMES:
Assessment of binocular far and intermediate visual acuity | 12 months
  Binocular far and intermediate visual acuity in logMar will be measured at 4 metre and 70 cm distance using an ETDRS visual acuity chart
Assessment of halos | 12 months
  Extent of halos will be measured and analysed using the Aston halometer
Assessment of binocular contrast sensitivity | 12 months
  Binocular contrast sensitivity will be measured using the Optec Vision tester under mesopic and photopic conditions
Assessment of reading speed | 12 months
  Patients reading speed will be measured using the Salzburg Reading Desk

CONTACTS AND LOCATIONS:
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided